CLINICAL TRIAL: NCT05383001
Title: Randomized Phase II, Open-label Efficacy and Safety Study of Second-line Durvalumab Plus Tremelimumab Versus Platinum-based Chemotherapy Alone in Patients With NSCLC and First-line Checkpoint-inhibitor Therapy Followed by 2 Cycles of Platinum-based Chemotherapy (Re-Check)
Brief Title: Randomized Phase II, Open-label Efficacy and Safety Study of Second-line Durvalumab Plus Tremelimumab Versus Platinum-based Chemotherapy Alone in Patients With NSCLC and First-line Checkpoint-inhibitor Therapy (Re-Check)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was set-up in 2017, even though the protocol was adjusted, it was not possible to find suitable patients.
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-TRK-0221; 2017-003780-35 (EudraCT Number); ESR-17-12719 (Other Grant/Funding Number: AstraZeneca GmbH)
Record Dates: First submitted 2022-05-17; First posted 2022-05-19 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: tremelimumab /durvalumab (1 cycle), subsequently Durvalumab maintenance therapy (Experimental)
  Interventions: Drug: combination regimen tremelimumab /durvalumab
- Arm B: platinum-based chemotherapy (SoC) (Other)
  Interventions: Drug: platinum-based chemotherapy (SoC)

INTERVENTIONS:
Drug: combination regimen tremelimumab /durvalumab — Induction treatment: 2 cyles of Q3W second-line plantium-based chemotherapy according to standard of care: Cisplatin or carboplatin in combination with pemetrexed, paclitaxel, nab-paclitaxel, vinorelbine or gemcitabine
  Combination treatment:
  Durvalumab 1500 mg fixed dose plus tremelimumab 300 mg fixed bolus dose
  Maintenance Therapy:
  Durvalumab 1500 mg fixed dose Q4W up to 12 cycles within the study
  Arms: Arm A: tremelimumab /durvalumab (1 cycle), subsequently Durvalumab maintenance therapy
Drug: platinum-based chemotherapy (SoC) — Induction treatment: 2 cyles of Q3W second-line plantium-based chemotherapy according to standard of care: Cisplatin or carboplatin in combination with pemetrexed, paclitaxel, nab-paclitaxel, vinorelbine or gemcitabine
  Combination treatment:
  Continuation of second-line chemotherapy with 2-4 further cycles (Q3W) platinum-based combination therapy.
  Maintenance Therapy:
  Optional continued maintenance therapy with pemetrexed according to marketing authorization will be allowed for a maximum of 13 cycles.
  Arms: Arm B: platinum-based chemotherapy (SoC)

SUMMARY:
This is an open label, randomized, Phase II multicenter study designed to evaluate the safety and efficacy of two different second-line strategies: After failure of first line mono-immunotherapy with checkpoint inhibitors (anti-PD-1/PD-L1), and subsequent 2 cycles of standard of care platinum-based chemotherapy, 2 treatment arms will be compared: Arm A (Experimental Arm): After randomization, patients will receive a combination regimen featuring a single, priming dose of tremelimumab together with conventional durvalumab dosing. Durvalumab maintenance therapy will subsequently be continued as study treatment for up to 12 cycles.

Arm B: After randomization, patients will continue to receive another 2-4 cycles of platinum-based chemotherapy. Afterwards, patients will end treatment or receive maintenance pemetrexed therapy as per marketing authorization (depending on histology, maximum of 13 cycles) at the discretion of the investigator

DETAILED DESCRIPTION:
Patients without progression after two cycles of chemotherapy (induction treatment phase) will be randomized at a 1:1 ratio into one of 2 treatment arms (combination treatment phase). PD-L1 expression status will be evaluated based on available data. To better focus on patients with expected good clinical benefit from immunomodulating agents, only patients with checkpoint-inhibitor treatment as first-line monotherapy and a progression-free survival of at least 12 weeks will enter the study (at least two re-assessments after initiation of first-line treatment). Consequently, patients with disease progression as best response of first-line therapy cannot enter this study. Directly re-challenging patients with anti-PD-L1 and anti-CTLA agents after disease progression on checkpoint-inhibitor monotherapy will be avoided by the previous application of two cycles of platinum-based chemotherapy as induction treatment, which may also enhance the antigen release from tumor cells and may further support the subsequent immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Age >18 years at time of study entry
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Histologically or cytologically confirmed, stage IV NSCLC (per the Union Internationale contre le Cancer/American Joint Committee on Cancer staging system).
5. Indication for standard-of-care second line platinum-based chemotherapy, using cisplatin or carboplatin in combination with pemetrexed, paclitaxel, nab-paclitaxel, vinorelbine or gemcitabine
6. Life expectancy of > 12 weeks
7. Body weight > 30 kg
8. First-line mono-immunotherapy with checkpoint inhibitors (anti-PD1/PD-L1) with a best response of stable disease (SD) or better
9. Documented tumor PD-L1 expression status of ≥50%. Any existing data can be used.
10. First-line progression-free survival of at least 12 weeks after at least two re-assessments after initiation of first-line treatment.
11. Patients who have received prior neo-adjuvant, adjuvant chemotherapy, or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 6 months from initiation of first-line immunotherapy since the last adjuvant chemotherapy or chemoradiotherapy cycle.
12. Patients with a history of treated asymptomatic CNS metastases are eligible, provided they meet all of the following criteria:

    * No ongoing requirement for corticosteroids as therapy for CNS disease
    * No stereotactic radiation within 7 days or whole-brain radiation within 14 days prior to enrolment
    * No evidence of interim progression between the completion of CNS-directed therapy and the screening
    * Only supratentorial and cerebellar metastases allowed (i.e., no metastases to midbrain, pons, medulla or spinal cord)
13. No known sensitizing mutation in the EGFR gene or evidence of an ALK fusion oncogene.
14. Measurable disease, as defined by RECIST v1.1. Previously irradiated lesions can only be considered as measurable disease if disease progression has been unequivocally documented at that site since radiation.
15. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 3 days prior to enrolment:

    1. ANC 1500 cells/μL without granulocyte colony-stimulating factor support
    2. Lymphocyte count ≥ 500/μL
    3. Platelet count ≥ 100,000/μL without transfusion
    4. Hemoglobin ≥ 9.0 g/dL. Patients may be transfused to meet this criterion. Transfusions are allowed throughout the study.
    5. Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    6. AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
    7. Measured creatinine clearance (CL) >60 mL/min or calculated creatinine clearance CL>60 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24- hour urine collection for determination of creatinine clearance

Exclusion Criteria:

1. Use of immunosuppressive medication (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor [anti-TNF] agents) within 14 days prior to randomization. The following are exceptions to this criterion:

* Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be eligible after discussion with the study chair.
* The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
* Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
* Systemic corticosteroids at physiologic doses not exceeding 10 mg/day of prednisone or its equivalent
* Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).

Prior treatment with other immune-modulating agents (other than anti-PD-1/PD-L1) 3. Treatment with systemic immunostimulatory agents (including but not limited to IFNs, IL-2) within 4 weeks or five half-lives of the drug, whichever is longer, prior to randomization. Prior treatment with cancer vaccines is allowed.

4. Involvement in the planning and/or conduct of the study (applies to both sponsor staff and/or staff at the study site) 5. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study 6. Treatment with any other investigational agent or participation in another clinical study with therapeutic intent within 28 days prior to randomization 7. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy (including second line platinum-based chemotherapy) with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

• Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Chair.

* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Chair.

  8. Any toxicity that led to permanent discontinuation of prior immunotherapy. 9. A ≥ grade 4 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy.

  10. Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.

  11. History of allogenic organ transplantation. 12. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.

  13. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:
* Patients with vitiligo or alopecia
* Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Patients without active disease in the last 5 years may be included but only after consultation with the Study Chair
* Patients with celiac disease controlled by diet alone 14. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent 15. History of another primary malignancy except
* Malignancy treated with curative intent and with no known active disease ≥3 years prior to study enrolment and of low potential risk for recurrence
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated carcinoma in situ without evidence of disease 16. History of leptomeningeal carcinomatosis 17. History of active primary immunodeficiency 18. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. 19. Receipt of live or live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients should also not receive live or live attenuated vaccine for the pertinent time frames during and after treatment defined in the respective study drug's SmPC or IB.

  20. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

  21. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to a defined timepoint after last dose of treatment (see Section 7.1 for details) 22. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms); A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
PFS1 | 49 months
  Progression-free survival 1 using Investigator assessments according to RECIST 1.1, defined as the time from randomization in the study until objective tumor progression and do not include deaths

SECONDARY OUTCOMES:
PFS2 | 49 months
  Progression-free survival after initiation of second-line therapy
OS | 49 months
  Overall survival after initiation of second-line therapy
ORR | 49 months
  Objective response rate - Proportion of patients with CR or PR as best overall radiological tumor response counted from initiation of second-line treatment
Subgroup analysis | 49 months
  Objective response rate (best overall response) after randomization
DoR | 49 months
  Duration of response - Time from documentation of tumor response to disease progression
TFST | 49 months
  Time to first subsequent treatment - Time from initiation of second line treatment to initiation of third line treatment.
Tolerability and adverse events | 49 months
  Adverse events will be assessed by the type, seriousness, severity, and relatedness to treatment. A descriptive analysis of safety related laboratory parameters will complement the safety assessment.
QoL | 49 months
  Quality of Life measured with the EORTC QLQ-C30 (core questionnaire) and the QLQLC13 (lung cancer module)

CONTACTS AND LOCATIONS:
Overall Officials: Niels Reinmuth, Prof. Dr., Study Chair — Asklepios Fachkliniken München-Gauting, Thorakale Onkologie
Locations (1):
- Asklepios Fachkliniken München-Gauting, Gauting, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de/